CLINICAL TRIAL: NCT00274690
Title: A Multicenter, Randomised, Double-blind, Placebo-controlled, Parallel Group, Phase II Study to Evaluate the Safety and Efficacy of Oral Dosing With GW679769 (50 mg or 150 mg) for Three Consecutive Days When Administered With a Single Intravenous Dose of Ondansetron Hydrochloride for the Prevention of Post-operative Nausea and Vomiting and Post-discharge Nausea and Vomiting in Female Subjects With Known Risk Factors for Post-operative Nausea and Vomiting Who Are Undergoing Laparoscopic/Laparotomic Surgical Procedures Associated With an Increased Emetogenic Risk
Brief Title: Post-Operative Nausea And Vomiting Study In Female Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NKT102245
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Nausea and Vomiting; Nausea and Vomiting, Postoperative
Keywords: Neurokinin-1 Receptor Antagonist; GW679769; Post-operative Nausea; NK-1 Receptor Antagonist; PONV; Post-discharge Nausea and Vomiting; PDNV; Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769

SUMMARY:
The primary purpose of this study is to determine an effective dose of this NK-1 anti-emetic medication to prevent nausea and vomiting in females after surgery.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase II Study to Evaluate the Safety and Efficacy of Oral Dosing with GW679769 (50 mg or 150 mg) for Three Consecutive Days When Administered with a Single Intravenous Dose of Ondansetron Hydrochloride for the Prevention of Post-operative Nausea and Vomiting and Post-discharge Nausea and Vomiting in Female Subjects with Known Risk Factors for Post-operative Nausea and Vomiting Who are Undergoing Laparoscopic/Laparotomic Surgical Procedures Associated with an Increased Emetogenic Risk

ELIGIBILITY:
Inclusion Criteria:

* Known, specified risk factors for PONV (post operative nausea and vomiting)
* Undergoing gynecologic or gallbladder surgery.

Exclusion Criteria:

* pregnant or breastfeeding
* post-menopausal

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 435 (Actual)
Dates: Start 2005-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who achieve a complete response (defined as no vomiting, no retching, no rescue therapy, & no premature discontinuation from the study) during the first 72 hr evaluation period following the emergence from anesthesia. | 72 Hours

SECONDARY OUTCOMES:
The proportion of subjects who achieve a complete response during each subsequent 24-hr eval period (up to 120 hrs) following the emergence from anesthesia. | 120 Hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- United States (11):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Seattle, Washington
- Denmark (3):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Viborg
- Hong Kong (5):
  - GSK Investigational Site, Lai Chi Kok
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shamshuipo, Kowloon
  - GSK Investigational Site, Shatin, New Territories
  - GSK Investigational Site, Tuenmen
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szentes
- Israel (2):
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Tel Litwinsky
- Norway (3):
  - GSK Investigational Site, Gjettum
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Skien
- GSK Investigational Site, Manila, Philippines
- Slovenia (3):
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Novo Mesto
  - GSK Investigational Site, Slovenj Gradec
- Spain (4):
  - GSK Investigational Site, Badalona(Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (4):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Livingston, West Lothian
  - GSK Investigational Site, Hull